CLINICAL TRIAL: NCT04348578
Title: Effect of QMix 2-in-1 as Final Irrigation Protocol on Periapical Healing After Single-visit Root Canal Treatment: a Randomized Controlled Trial
Brief Title: Effect of QMix 2in1 as Final Irrigation Protocol on Periapical Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cemre Sapmaz Uçan, Research Asistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDH-2017-8165
Record Dates: First submitted 2020-04-08; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Periapical Diseases
Keywords: QMix 2-in-1; Sodium hypochlorite; Chlorhexidine; Treatment outcome; Radiographic healing
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (No Intervention): The root canal was prepared using the WaveOne Gold file reciprocation system with VDW Silver motor. WaveOne Gold #25 (0.07) file was used for instrumentation. For larger canals, #35 (0.06) and #45 (0.05) files were used after the #25 file. During instrumentation procedure, irrigation was applied with 5mL 2.5% NaOCl using a side-vented needles. The final irrigation was applied with 5mL NaOCl and 5mL sterile saline in the control group.The root canals were dried with sterile paper points and were filled with gutta-percha and AH Plus sealer with the cold lateral condensation method and the entry cavity was restored with composite. All treatments were performed following a standardized procedure by one operator. After completion of the root canal treatment, periapical radiographs were taken using the paralleling technique. All the patients were called for follow-up examination at 12 months, and were examined radiographically.
- QMix 2in1 (Experimental): The root canal was prepared using the WaveOne Gold file reciprocation system with VDW Silver motor. WaveOne Gold #25 (0.07) file was used for instrumentation. For larger canals, #35 (0.06) and #45 (0.05) files were used after the #25 file. During instrumentation procedure, irrigation was applied with 5mL 2.5% NaOCl using a side-vented needles. The final irrigation was applied with 5mL Mix 2in1 and 5mL sterile saline in the experimental group.
  Interventions: Other: QMix 2in1

INTERVENTIONS:
Other: QMix 2in1 — In QMix 2in1 group root canals were irrigated with Mix as a final irrigation.
  Arms: QMix 2in1

SUMMARY:
Aim: To compare the 12-month radiographic outcome of root canal treatment with and without the additional use of QMix 2-in-1 (Dentsply Tulsa, Maillefer, Ballaigues, Switzerland) irrigation solution.

Methodology: The study included 60 single-rooted teeth with periapical radiolucency of 60 patients, randomized into two groups using randomized block design with block sizes of 10 patients in each. Root canals were prepared with WaveOne Gold files (Dentsply Sirona, Maillefer, Ballaigues, Switzerland) and irrigation was performed with 5 mL 2.5% sodium hypochlorite (NaOCl) using side-vented needles during instrumentation. The final irrigation protocol was performed using 5 mL 2.5% NaOCl (n= 30) or 5 ml QMix 2-in-1 (n=30). Then the root canals were irrigated with 5 mL of distilled water and filled with gutta-percha and AH Plus sealer (Dentsply Sirona), using the cold lateral compaction technique. The patients were recalled after 12 months and evaluated radiographically according to perapical index (PAI) scores. Pre and post-treatment PAI scores were compared and teeth were considered 'healthy' (PAI ≤ 2) or 'diseased' (PAI ≥ 3). The Mann Whitney U test was used to compare the differences between the post-operative and follow-up images of the treatment groups. The Wilcoxon signed rank test was applied to examine the changes in PAI score from baseline to the follow-up evaluation in each group.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted to evaluate radiographic periapical repair after endodontic treatment using QMix 2-in-1 (Dentsply Tulsa, Maillefer, Ballaigues, Switzerland) and NaOCl irrigation in single-rooted teeth with apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* necrotic, single root teeth with a periapical lesion (2>PAI>5)

Exclusion Criteria:

* pregnant
* had used antibiotics within the previous week
* allergy to local anesthetic agents
* history of intolerance to non-steroidal anti-inflammatory drugs
* had uncontrolled hypertension, uncontrolled diabetes mellitus, chronic renal failure, hematological disease, or had received or were receiving radiotherapy and periodontal bone loss (visualized radiographically)
* open tooth apex

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Radiographic healing after 12 months follow-up. | Time frame is 12 months for this study. Each patient will recall for an appointment and the status of the tooth will evaluate radiographically.
  After the completion of treatment of both control and QMix 2in1 group, the status of periapical healing was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Yoldaş, Professor, Study Director — University of Cukurova, Faculty of Dentistry, Vice-Dean
Locations (1):
- Cukurova University, Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbaszadegan A, Nabavizadeh M, Hoseini Yekani A, Khayat A. Comparison of Endodontic Treatment Results Yielded from Using Normal Saline with IKI Final Rinse or NaOCl Irrigation: A 30-Month Follow-up Study. Iran Endod J. 2013 Fall;8(4):171-6. Epub 2013 Oct 7. PMID 24171024
- [Result] Holland R, Gomes JE Filho, Cintra LTA, Queiroz IOA, Estrela C. Factors affecting the periapical healing process of endodontically treated teeth. J Appl Oral Sci. 2017 Sep-Oct;25(5):465-476. doi: 10.1590/1678-7757-2016-0464. PMID 29069143
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- [Result] Pai S, Thomas MS. The effect of QMix, an experimental antibacterial root canal irrigant, on removal of canal wall smear layer and debris. J Endod. 2011 Jun;37(6):741; author reply 741-3. doi: 10.1016/j.joen.2011.04.006. Epub 2011 May 6. No abstract available. PMID 21787479
- [Result] Chandrasekhar V, Amulya V, Rani VS, Prakash TJ, Ranjani AS, Gayathri Ch. Evaluation of biocompatibility of a new root canal irrigant Q Mix 2 in 1- An in vivo study. J Conserv Dent. 2013 Jan;16(1):36-40. doi: 10.4103/0972-0707.105296. PMID 23349574